CLINICAL TRIAL: NCT04641260
Title: A Phase 1 Crossover Study to Investigate the Effect of Food on the Pharmacokinetics of Fezolinetant in Healthy Female Participants
Brief Title: A Study to Assess the Effect of Food With Fezolinetant in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2693-CL-0012
Record Dates: First submitted 2020-11-20; First posted 2020-11-23 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics of Fezolinetant; Effect of Food; ESN364
MeSH Terms: interventions — fezolinetant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fezolinetant: Fed State then Fasted State (Experimental): Participants will receive a single oral dose of fezolinetant in fed state on day 1 of study period 1. After a washout of 5 days the participants will receive a single oral dose of fezolinetant in fasted state on day 1 of study period 2.
  Interventions: Drug: Fezolinetant
- Fezolinetant: Fasted State then Fed State (Experimental): Participants will receive a single oral dose of fezolinetant in fasted state on day 1 of study period 1. After a washout of 5 days the participants will receive a single oral dose of fezolinetant in fed state on day 1 of study period 2.
  Interventions: Drug: Fezolinetant

INTERVENTIONS:
Drug: Fezolinetant — Oral
  Other Names: ESN364

SUMMARY:
The purpose of this study is to evaluate the effect of food on the pharmacokinetics of a single oral dose of fezolinetant under fasted and fed conditions in healthy female participants. The study will also evaluate the safety and tolerability of a single oral dose of fezolinetant under fasted and fed conditions in healthy female participants.

DETAILED DESCRIPTION:
Each participant will participate in 2 treatment periods separated by a washout of at least 5 days between investigational product (IP) administration in each period. Participants will be admitted to the clinical unit on day -1 of period 1 and will be in clinical unit for periods 1 and 2. On day 1 of each period, participants will receive fezolinetant followed by a 72-hour blood sampling period. The study will be completed with an end-of-study visit (ESV) which will take place 5 to 9 days after the 72-hour blood sampling period in period 2 or at the time of early discontinuation from the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a body mass index (BMI) range of 18.5 to 34.0 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance for at least 30 days prior to day -1 of period 1 through at least 30 days after final IP administration
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for 30 days after final IP administration.
* Female participant must not donate ova starting at first dose of IP and throughout the study period and for 30 days after final IP administration.
* Participant agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has any condition which makes the participant unsuitable for study participation.
* Female participant who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Participant has a known or suspected hypersensitivity to fezolinetant or any components of the formulation used.
* Participant has had previous exposure with fezolinetant.
* Participant has any of the liver function tests (alkaline phosphatase [ALP], alanine aminotransferase [ALT], aspartate aminotransferase [AST] and total bilirubin [TBL]) > 1.5 × the upper limit of normal (ULN) on day -1 of period 1. In such a case, the assessment may be repeated once.
* Participant has creatinine level outside normal limits on day -1 of period 1. In such a case, the assessment may be repeated once.
* Participant has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to first IP administration.
* Participant has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1 of period 1.
* Participant has any clinically significant abnormality following the physical examination, ECG and protocol-defined clinical laboratory tests at screening or on day -1 of period 1.
* Participant has a mean pulse of < 45 or > 90 bpm or systolic blood pressure ≥ 130 millimeters of mercury (mmHg) or diastolic blood pressure ≥ 80 mmHg based on the average of 3 readings. These 3 readings must occur on at least 2 different occasions during the screening period or on day -1 of period 1. Repeat measurements will not be taken during screening, but may be taken on day -1 of period 1.
* Participant has a mean corrected QT interval using Fridericia's formula (QTcF) of > 470 msec on day -1 of period 1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Participant has used any prescribed or nonprescribed drugs (including vitamins, oral contraceptives or hormone replacement therapy [HRT] and natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to first IP administration except for occasional use of acetaminophen (up to 2 g/day) and topical dermatological products (including corticosteroid products).
* Participant has smoked, used tobacco-containing products and nicotine or nicotine-containing products (e.g., electronic vapes) within 6 months prior to screening or the participant tests positive for cotinine at screening or on day -1 of period 1.
* Participant has a history of consuming > 7 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the participant tests positive for alcohol at screening or on day -1 of period 1.
* Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 of period 1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or on day -1 of period 1.
* Participant has used any inducer of cytochrome P450 (CYP) 1A2 in the 3 months prior or inhibitors of CYP 1A2 in the 2 weeks or 5 half-lives of the inhibitor, whichever is longer, prior to day -1 of period 1.
* Participant has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day 1 and/or received a transfusion of any blood or blood products within 60 days.
* Participant has a positive serology test for hepatitis A virus antibodies (immunoglobulin M), hepatitis B core antibodies, hepatitis B surface antigen, hepatitis C virus antibodies or antibodies to human immunodeficiency virus type 1 and/or type 2 at screening.
* Participant is an employee of Astellas, the study-related contract research organizations (CROs) or the clinical unit.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of fezolinetant in plasma: Area under the concentration-time Curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf) | up to Day 4 in each study period.
  AUCinf will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: Area under the concentration-time curve (AUC) from the time of dosing to the last measurable concentration (AUClast) | up to Day 4 in each study period.
  AUClast will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: Maximum concentration (Cmax) | up to Day 4 in each study period.
  Cmax will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: Time of maximum concentration (Tmax) | up to Day 4 in each study period.
  Tmax will be recorded from the PK plasma samples collected.

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | up to Day 18
  An AE is any untoward medical occurrence in a participant administered an IP, whether or not considered related to the IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP. This includes events related to the comparator and events related to the (study) procedures.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | up to Day 18
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or adverse events (AEs) | up to Day 18
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | up to Day 18
  Number of participants with potentially clinically significant electrocardiogram (ECG) values.

CONTACTS AND LOCATIONS:
Overall Officials: Executive Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Parexel, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.